CLINICAL TRIAL: NCT00579852
Title: A Prospective Trial to Assess the Variability of Uni-Dimensional, Bi-Dimensional, and Volumetric CT Scan Measurement of Non-Small Cell Lung Cancer Tumors
Brief Title: Assess the Variability of Uni-Dimensional, Bi-Dimensional, and Volumetric CT Scan Measurement of Non-Small Cell Lung Cancer Tumors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Mark Kris, MD, Memorial Sloan-Kettering Cancre Center
Other Study IDs: 06-149
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Lung Cancer; Non Small Cell
Keywords: Lung
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: Patients with NSCLC undergoing non-contrast CT scan of the chest will have a second, high resolution, non-contrast CT scan of the chest performed on the same day.
  Interventions: Procedure: CT Scan

INTERVENTIONS:
Procedure: CT Scan — Patients with NSCLC undergoing non-contrast CT scan of the chest will have a second, high resolution, non-contrast CT scan of the chest performed on the same day. The scans will be performed on the same CT scanner, generally within 30 minutes. Unidimensional, bi-dimensional, and volume measurements for the primary NSCLC lesion will be determined on both scans and the values compared. After completing the second scan, the patient will have completed participation in the protocol.

SUMMARY:
The purpose of this study is to compare the results of two CT scans of the chest performed within minutes of each other. We will compare several different measurements of lung cancer tumors. This study will help show whether we can get accurate results when we compare measurements on different CT scans. This information is important for patients with cancer, who often have more than one CT scan during their treatment.

DETAILED DESCRIPTION:
Standard criteria for tumor response assessment have used uni-dimensional or bi-dimensional measurements as a surrogate for volume determination. Modern CT scan techniques, in combination with algorithms developed at MSKCC, allow the calculation of tumor volume. This protocol is designed to evaluate the reproducibility of the calculated volume of pulmonary masses on separate CT scans obtained on the same day in patients with non-small cell lung cancer (NSCLC). Patients with NSCLC undergoing non-contrast CT scan of the chest will have a second, non-contrast CT scan of the chest performed. Uni-dimensional, bi-dimensional, and volume measurements for the primary NSCLC lesion will be determined on both scans and the values compared.

ELIGIBILITY:
Inclusion Criteria:

* Have pathologically confirmed non-small cell lung cancer
* Have measurable primary pulmonary tumors ≥ 1cm
* Have plans for a clinically indicated non-contrast CT scan of the chest
* All patients must be ≥ 18 years old

Exclusion Criteria:

* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thoracic Oncology Service at MSKCC clinic.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2006-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the reproducibility of calculated volume of pulmonary masses on separate CT scans obtained on the same day in patients with NSCLC | same day, within 30 minutes

SECONDARY OUTCOMES:
To evaluate the reproducibility of bidimensional and unidimensional measurement of pulmonary masses on separate CT scans obtained on the same day in patients with NSCLC | same day, within 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Oxnard GR, Zhao B, Sima CS, Ginsberg MS, James LP, Lefkowitz RA, Guo P, Kris MG, Schwartz LH, Riely GJ. Variability of lung tumor measurements on repeat computed tomography scans taken within 15 minutes. J Clin Oncol. 2011 Aug 10;29(23):3114-9. doi: 10.1200/JCO.2010.33.7071. Epub 2011 Jul 5. PMID 21730273
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org